CLINICAL TRIAL: NCT04723641
Title: Effect of Functional Strength Training From Plantigrade Foot Position on Motor Performance in Children With Diplegia
Brief Title: Effect of Functional Training on Motor Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, hanaa mohsen, lecturer,department of physical therapy for pediatrics and pediatric surgery, badr university in cairo, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hana 5
Record Dates: First submitted 2021-01-19; First posted 2021-01-26 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Diplegia

STUDY DESIGN:
Intervention Model Description: intervention group received progressive resistive functional strength training from plantigrade foot position conducted for one hour, 3 days/week. The therapist will replace the conventional physical therapy with the progressive resistive functional strength training, when this is consistent with the objectives of the strength training.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STUDY GROUP (Experimental): they received progressive resistive functional strength training from plantigrade foot position conducted for one hour, 3 days/week. The therapist will replace the conventional physical therapy with the progressive resistive functional strength training, when this is consistent with the objectives of the strength training.
  Interventions: Other: functional training exercises
- control group (No Intervention): received a designed physical therapy program

INTERVENTIONS:
Other: functional training exercises — progressive resistive functional strength training from plantigrade foot position conducted for one hour, 3 days/week. The therapist will replace the conventional physical therapy with the progressive resistive functional strength training, when this is consistent with the objectives of the strength training.
  Arms: STUDY GROUP

SUMMARY:
The functional strength training is mainly dealt with anti-gravity muscles and aiming at maximal carry over in day to day activities. The functional strength training can be given using resistance and it may be gravity, body weight, resistance bands and free weights. The exercises are specific to the muscle or muscle groups recruited during the functional activities

ELIGIBILITY:
Inclusion Criteria:

1. Age ranged from 7 to 10 years old.
2. The degree of spasticity ranged from grade 1 to 2 hypertonia according to Modified Ashwarth Scale (MAS)
3. Level II and III on GMFCS-ER
4. They were able to understand and follow verbal instructions

Exclusion Criteria:

* 1- visual or auditory problems. 2- Orthopedic surgery in the lower limb in the last 12 months before the study. 3- Fixed deformities in joints and bones of lower limbs. 4- Botox injection in the last six months before the study. 5- Children with any special medications affecting muscle functions (anti-spastic drugs).

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Gross motor functional measurement | pre and after 3 months of intervention,, the higer score will represent the improvement
  The GMFM is a standardized observational scale designed and validated to measure change in gross motor function over time in children with CP.

SECONDARY OUTCOMES:
Isometric muscle strength measurements | pre and after 3 months of intervention,, increase in muscle will represent the improvement
  The gold standard for evaluating isometric muscle strength is the portable dynamometer. This is an easy-to-use, sensitive device for detecting muscular action and for performing objective, valid, and reliable measurements in several populations

CONTACTS AND LOCATIONS:
Locations (1):
- Hanaa, Cairo, Egypt